CLINICAL TRIAL: NCT04270890
Title: Analysis of an Abdominal Compression Device to Reduce Respiratory Motion of Lower Thorax and Abdominal Tumours
Brief Title: Investigation of an Abdominal Compression Device
Acronym: ACE02
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Clatterbridge Cancer Centre NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CO966
Record Dates: First submitted 2020-02-11; First posted 2020-02-17 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-02

CONDITIONS: Cancer, Lung; Cancer of Stomach
Keywords: ablative stereotactic radiotherapy,; lung cancer; compression device
MeSH Terms: conditions — Lung Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study participants (Experimental): Patients will be dual scanned; one with 4D-CT in free-breathing and one wearing the compression belt.Organ motion will then be quantified using Eclipse. This facilitates a direct comparison to determine the efficacy of the compression belt. Patients with reduction in organ motion will be treated wearing the abdominal compression belt. The alignment scale will be recorded to facilitate accurate placement each fraction. The belt will be inflated to a tolerable level by the patient and recorded for consistency each fraction. The position of the belt will be referenced to the anterior and lateral tattoos to ensure accurate and consistent placement each fraction.
  Interventions: Device: Abdominal compression belt system

INTERVENTIONS:
Device: Abdominal compression belt system — The abdominal compression belt system is provided free of charge from CDR systems, Canada.
  The belt has specifically been chosen from other similar devices commercially available as it is independent of other immobilisation devices and can be used with the patient located within a full body vacbag as per current immobilisation position.

SUMMARY:
This study is applicable to patients undergoing lower lung or abdomen stereotactic ablative body radiotherapy (SABR) treatment. The purpose of the ACE 01 study is to identify if, the volume of healthy tissue within the treatment area and therefore subsequent side effects, can be reduced by using a commercially available abdominal compression device to minimise breathing related movement. The secondary aim will be to assess patient compliance and comfort of thedevice. This will be assessed by asking the patient to complete a 'patient comfort questionnaire'. In addition the radiographers will be asked to complete a 'satisfaction questionnaire' to determine ease and reproducibility of use.

DETAILED DESCRIPTION:
Stereotactic ablative body radiotherapy (SABR) offers the ability to deliver a high dose of radiotherapy accurately to small tumours. It is an established, effective, non-invasive treatment option for early lung cancers as an alternative to surgery and in the treatment of limited spread of cancer (called oligo-metastatic disease) in the context of clinical trials (CORE, SARON, ABC-07 etc.). In order to deliver a high dose of radiation without damaging the surrounding structures, an accurate map of the tumour and the surrounding organs and their relationship to each other when moving (for e.g. during breathing) is important. This is usually achieved by getting a radiotherapy treatment planning 4 dimensional CT scan (4D-CT). When either the tumour or organ around them (like the lung) are moving excessively it becomes difficult to target the radiation beams and often the only solution is to treat a larger volume which covers the extent of the movement. Treating larger volumes often leads to more toxicity to the surrounding tissues.Therefore managing motion is critical to increasing tumour control probability (TCP) and reducing normal tissue complication probability (NTCP). In this context, the question of reducing the movement caused by breathing, of tumours in the lower lung and upper abdomen (like the liver, adrenals, kidney etc) is an area of intense interest. Various technical and physical methods exist to help improve motion management in patients under going radiotherapy. By limiting the movement, the target volume is smaller and this enables treatment of the tumour to high doses with lesser toxicity as some of the toxicity of radiotherapy is proportionate to the volume treated i.e. lower the volume of treatment lesser the risk of toxicity.

Abdominal compression is one such method and is well accepted to be beneficial in reducing tumour motion.

However, many of the previous studies require expensive and resource intensive immobilisation devices, costing, in many cases in excess of £10,000. This study will investigate the use of an independent compression device which can be used with any existing immobilisation system and costs in the region of £1,500. If proven to be beneficial this will allow many smaller centres or centres with budget limitations to also achieve the benefits of abdominal compression without extensive resource and cost requirements.

ELIGIBILITY:
Inclusion Criteria:

* • Radiological or Histologically confirmed lower lobe lung cancer or histologically confirmed metastatic of primary cancer in abdominal organs including liver, pancreas, adrenal which meets criteria for SABR treatment.

  * Aged 18 years or over
  * Capacity to understand research proposal and give informed consent

Exclusion Criteria:

* Tumour sites excluding those previously defined
* Rib metastases
* Stoma if situated underneath belt
* Patients unable to tolerate the abdominal compression belt
* Patients with existing abdominal aortic aneurysm (AAA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-06-21 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
To measure change in treatment volume between freebreathing and abdominal compression scans | 2 years
  Organ motion will then be quantified using Eclipse. This facilitates a direct comparison to determine the efficacy of the compression belt. Patients with reduction in organ motion will be treated wearing the abdominal compression belt. The alignment scale will be recorded to facilitate accurate placement each fraction.
  compression belt

SECONDARY OUTCOMES:
Reported patient feedback regarding device comfort and compliance of use. | 2 years
  The comfort of the device in clinical use will be measured by using a questionnaire that the patient will be asked to complete at initial scanning and then on two subsequent treatments. The results will be collated and analysed to qualitatively measure patient comfort and use of the device

CONTACTS AND LOCATIONS:
Overall Officials: Anoop Haridass, MD, Principal Investigator — Clatterbridge Cancer Centre
Locations (1):
- Clatterbridge Cancer Centre NHS Foundation Trust, Bebington, United Kingdom

IPD SHARING:
Plan to Share IPD: No